Service Dog Training Program for Military Veterans With PTSD NCT03777020 05-30-2023

Service Dog Training Program for Military Veterans With PTSD NCT03777020 10-10-22

### **Protocol**

This RCT will gather data from 60 veterans with Post-traumatic stress disorder (PTSD) and 30 service dogs (SDs) in training. Veterans will be recruited and screened for eligibility according to Warrior Canine Connection (WCC) inclusion criteria Humans: 1) military veteran; 2) diagnosis of PTSD; 3) able to give informed consent; and 4) able to understand English. Human Exclusion Criteria: 1) fear of dogs; 2) allergy to pet dander; 3) active substance abuse; 4) active psychosis, or 5) history of animal abuse. Dog Inclusion Criteria: 1) non-aggressive demeanor as evaluated by WCC protocols for evaluating animal temperament; 2) cleared by veterinarian; and 3) up-to date immunizations. Dog Exclusion Criteria: 1) medical holds.

Recruitment/Screening:. Recruitment will be via media attention, flyers, social media, and word of mouth.

<u>Procedures:</u> Veterans interested in the participating in the study will be prescreened by a research team member(RTM) for eligibility. Eligible veterans will be invited to participate. If veterans agree to participate after their questions are answered. They will be consented verbally, randomized, and scheduled for their first session with the location dependent on the arm. After informed consent is signed, baseline data will be obtained in an outdoor area at WCC [service dog training program(SDTP) arm] or at another meeting place near the participant's home [wait list control intervention((WLCI) arm].

<u>Randomization:</u> Participants will be block randomized, according to gender, into the SDTP or WLCI. Group assignments will be generated by a computerized random number table and envelopes will be opened after verbal informed consent. Participants will continue existing therapies and begin any for which they are referred while in the study.

### **Interventions:**

<u>SDTP-Intervention (human)</u>: Veterans randomized to the SDTP will be paired with an experienced WCC Mission Based Trauma Recovery (MBTR)-Trainer (MBRT-T) and a SD. One hour training modules will be scheduled once a week for 8 weeks. Participants will come to WCC for all the weekly training modules. The MBTR-T will deliver the prescribed SDTP modules created by WCC. Each session will be fully supervised by a WCC MBTR-T to address any concerns or safety issues that may arise.

<u>Waitlist Control Intervention (WLCI)</u>: Veterans randomized to WLCI will participate in one hour online SD training modules (<a href="https://e-trainingfordogs.com">https://e-trainingfordogs.com</a></u>) scheduled once a week for 8 weeks but not interact with service dogs. The online training modules are delivered by experienced SD trainers and will employ parallel content to the WCC SDTP. Participants will participate from their homes or at a location of their choice in online training modules.

Outcome Assessment: In both groups, human's biological [e.g. salivary and heart rate variability (HRV)] markers except telomere length (TL) will be assessed in weeks 1, 4, and 8. TL will be assessed at weeks 1 and 8. Scales for and psychosocial data will be completed prior to session 1 and after sessions 4 and 8. HRV will be recorded in the human participants during SDTP sessions and for 30 minutes after sessions.

<u>Assessment</u>: Human Demographics and Characteristics Questionnaire will collect demographic/descriptive data on the human participants, such as gender, age, race, ethnicity, marital status, educational level, living arrangements, military history and pet ownership history. The order of the questionnaires will be randomized to minimize order effects. A dog demographics and characteristics questionnaire will collect demographic/descriptive data including dog's name, WCC dog trainer's name, gender, age, breed, and weight. Additionally, a photo will be taken to illustrate size and face.

# Aim 1 Outcome Assessment:

**Primary outcome:** <u>PTSDSS</u> will be assessed with the PTSD Checklist for DSM-5 (PCL-5), a 20-item scale.<sup>70</sup>.<sup>71</sup>

### **Secondary outcomes:**

- a) Stress markers will be assessed with salivary cortisol, α- amylase, and HRV, and the perceived stress scale. Heart <u>rate variability (HRV)</u> of veterans will be measured with a Polar H7 heart rate sensor worn around the chest and matching Polar V800 GPS Sports Watch worn around a wrist to save data from the heart rate sensor and download it for analysis. Perceived stress (PS) will be assessed with the Patient-Reported Outcomes Measurement Information System (PROMIS) Perceived Stress Fixed Form v2.0 (PROMIS, PS).<sup>72,73</sup> and
- b) Psychosocial health related to PTSD will be assessed with well validated scales, including PROMIS measures: Positive Affect-Short Form 15 (PA 15a), <sup>75</sup> PROMIS Satisfaction with Social Roles and Activities (SSRA) Short Form 4a (PROMIS-SSRA), <sup>80,81</sup> PROMIS Short Form v1.0- Satisfaction with Participation in Discretionary Social Activities- Short Form 7a (PROMIS SPDSA), <sup>82,83</sup> PROMIS Companionship Short Form 4a (PROMIS-C), <sup>84,85</sup> PROMIS Depression Short-Form 8a, <sup>87</sup> and the PROMIS Anxiety Short-Form 8a. <sup>88</sup> <u>Suicide ideation</u> (SI) will be assessed with the Beck Scale for Suicide Ideation. <sup>89</sup> Quality of life will be assessed with the Veterans RAND 12-Item Healthy Survey, <sup>76</sup> Resilience will be assessed with the Connor-Davidson Resilience Scale (CD-RISC-10), <sup>78</sup> and Quality of an individual's relationships will be assessed with the Relationship Scale Questionnaire (RSQ). <sup>79</sup>
- c) The exploratory outcome: cellular aging will be assessed by obtaining absolute telomere length analysis.<sup>90</sup>

<u>Aim 2 Outcome Assessment</u>: Dog HRV, is a reliable measure of stress levels.<sup>59,91</sup> will be measured with the PetPace Collar (http://petpace.com). This non-invasive, monitor wirelessly tracks the dog's HRV and a range of physical and behavioral parameters.

<u>Aim 3 Outcome Assessment</u>: Participant attendance and participation in each session will be recorded by the SD trainers. The SD trainers also keep extensive notes on the interactions between the veterans and the dogs. Documentation of unintended consequences such as aggressive behavior (on either part), allergic reactions, fearful behavior (on either part). These logs will be used to assess participation in the SDTP. Exit phone interviews will be used to obtain veterans' perceptions of the SDTP and their outcomes.

## **Data Analysis Plan**

<u>Human Data</u>: Before analyses, data will be cleaned and illustrated graphically. Summary statistics will be calculated, assumptions examined, and transformations applied as needed. Demographics and baseline characteristics (e.g., PTSDSS, gender) will be compared between the SDTP and WLCI groups, and the relevant variables considered as covariates for multivariable longitudinal analyses. SPSS 25 will be used for all analyses. Significance for rejecting the null is set at  $p \le .05$ , Bonferonni sequential corrections will be used for multiple comparisons. The intent-to-treat approach will guide hypothesis testing. Separate sets of analyses are conducted for each outcome.

**H1:** Participants in the SDTP (n = 30) will demonstrate significantly greater improvement in outcomes from week 1 to weeks 4 and 8 than the WLCI (n = 30) in: a) PTSD symptom severity; b) stress markers (decreased cortisol,  $\alpha$ -amylase, perceived stress; increased IgA, HRV); c) psychosocial health (increased positive affect, QOL, resilience, and relationships with friends and family, satisfaction with social activities and roles, companionship and decreased depression, anxiety, and suicide ideation); and d) exploratory stress marker cellular aging [increased TL, from weeks 1 to 8 only).

Linear mixed models (LMMs) with random intercepts (participant as a random variable) will be used to assess differences in changes in each outcome between the SDTP and WLCI participants, accounting for the correlation with the repeated measurements of each participant, and using all available data. Fixed effects will include group (SDTP or WLCI), week (1, 4 and 8), and their interaction, as well as the relevant covariates. The hypothesized effect of the intervention will be tested with the week by group interaction. Interactions of covariates (e.g. gender and age) with the group and time will be explored to provide information about their influence and for preliminary data to justify formal evaluation (with adequate power) in future studies. The multi-modal assessment in this study will provide the opportunity to explore characteristics that predict benefits.

<u>Dog data:</u> For analyses of data from dogs, demographics and baseline characteristics (e.g., size, gender, age), will be computed. The distributional characteristics of HRV (e.g., normality, outliers and missing) will be explored. Appropriate steps will be used as needed to ensure that applicable assumptions are met. Descriptive statistics will be computed for HRV by week and period (pre, during, and post).

**H2:** Dogs who participate in the SDTP will not experience increases in stress (decreases in HRV) from the 30 minutes before, to during, and after SDTP sessions. LMMs with random intercepts (dog as a random variable)

will be used to assess the significance of changes between the three periods, accounting for the correlation within the repeated measurements. Fixed effects will include period [pre, during, post SDTP session] and week (1, 4, 8). The hypothesized effect of the SDTP will be tested by evaluating the contribution of period to HRV. Interactions of dog covariates (e.g., dog gender and age) with period will explored to evaluate their potential influence and for exploring a need for evaluation of their roles.

**H3:** Dogs who participate in the SDTP will not experience increases in stress (decreases in HRV) over 8 weeks of the SDTP. The hypothesized effect of the intervention will be tested by evaluating contribution of week to HRV based on the LMM used for aim 2. Interactions of dog covariates (e.g. gender, age) with week will be explored to provide information about their potential influence to inform development of future studies. Feasibility data: Descriptive statistics will be calculated for number of sessions attended, rates of completion, drop out adverse events, and follow up questions, etc. Effect size estimates will be calculated for each veteran outcome and for dog HRV. They will enhance sample size calculations for a future multi-program RTC. **Missing Data**. While complete data are ideal and we will make considerable effort to obtain them, some missingness is likely. Randomness of missingness will be tested. If there is excessive or differential attrition across groups or informative missingness, we will apply sensitivity analysis, such as pattern mixture models for longitudinal data. If the results differ, we will report both.

#### References

- 1. Krause-Parello CA, Sarni S, Padden E. Military veterans and canine assistance for post-traumatic stress disorder: A narrative review. *Nurse Educ Today*. 2016;47:43-50. doi:10.1016/j.nedt.2016.04.020.
- 2. Bureau USC. FFF: Veterans Day 2017: Nov. 11. 2017.
- 3. Grieger TA, Cozza SJ, Ursano RJ, et al. Posttraumatic stress disorder and depression in battle-injured soldiers. *Am J Psychiatry*. 2006;163(10):1777-1783. doi:10.1176/ajp.2006.163.10.1777.
- 4. Sareen J, Cox BJ, Stein MB, Afifo TO, Fleet C, Asumundson GJ. Physical and mental comorbidity, disability, and suicidal behavior associated with post-traumatic stress disorder in a large community sample. *Psychosom Med.* 2007;63(3):242-248. doi:10.1097/PSY.0b013e31803146d8.
- 5. Besser A, Neria Y, Haynes M. Adult attachment, perceived stress, and PTSD among civilians exposed to ongoing terrorist attacks in Southern Israel. *Pers Individ Dif.* 2009;47(8):851-857. doi:10.1016/j.paid.2009.07.003.
- 6. Amstadter A. Emotion regulation and anxiety disorders. *J Anxiety Disord*. 2008;22(2):211-221. doi:10.1016/j.janxdis.2007.02.004.
- 7. Stellman JM, Smith RP, Katz CL, et al. Enduring mental health morbidity and social function impairment in world trade center rescue, recovery, and cleanup workers: The psychological dimension of an environmental health disaster. *Env Heal Perspect*. 2008;116(9):1248-1253. doi:10.1289/ehp.11164.
- 8. Davidson JR, Connor KM. Management of posttraumatic stress disorder: Diagnostic and therapeutic issues. *J Clin Psychiatry*. 1999;60(Suppl 18):33-38.
- 9. Tuerk PW, Yoder M, Grubaugh A, Myrick H, Hamner M, Acierno R. Prolonged exposure therapy for combat-related posttraumatic stress disorder: An examination of treatment effectiveness for veterans of the wars in Afghanistan and Iraq. *J Anxiety Disord*. 2011;25(3):397-403. doi:10.1016/j.janxdis.2010.11.002.
- 10. Shalev AY, Bonne O, Eth S. Treatment of posttraumatic stress disorder: A review. *Psychosom Med.* 1996;58(2):165-182.
- 11. Bradley R, Greene J, Russ E, Dutra L, Westen D. A multidimensional meta-analysis of psychotherapy for PTSD. *Am J Psychiatry*. 2005;162(2):214-227. doi:10.1176/appi.ajp.162.2.214.
- 12. Richardson JD, Contractor AA, Armour C, St Cyr K, Elhai JD, Sareen J. Predictors of long-term treatment outcome in combat and peacekeeping veterans with military-related PTSD. *J Clin Psychiatry*. 2014;75(11):e1299-305. doi:10.4088/JCP.13m08796.
- 13. Lancaster CL, Teeters JB, Gros DF, Back SE. Posttraumatic stress disorder: Overview of evidence-based assessment and treatment. *J Clin Med.* 2016;5(11):105. doi:10.3390/jcm5110105.
- 14. Congressional Budget Office. *The Veterans Health Administration's Treatment of PTSD and Traumatic Brain Injury among Recent Combat Veterans.*; 2012. https://www.cbo.gov/sites/default/files/112th-congress-2011-2012/reports/02-09-PTSD\_0.pdf.
- 15. Walsh PG, Mertin PG. The training of pets as therapy dogs in women's prison: A pilot study. *Anthrozoos*. 1994;7(2):124-128. doi:10.2752/089279394787002014.
- 16. Tull MT, Barrett HM, McMillan ES, Roemer L. A Preliminary Investigation of the Relationship between emotion regulation difficulties and posttraumatic stress symptoms. *Behav Ther.* 2007;38(3):303-313. doi:10.1016/j.beth.2006.10.001.
- 17. Institute of Medicine. Treatment for Posttraumatic Stress Disorder in Military and Veteran Populations: Final Assessment. Washington, DC; 2014. http://www.nationalacademies.org/hmd/~/media/Files/Report Files/2014/PTSD-II/PTSD-II-RB.pdf.
- 18. National Center for PTSD. Meditation-based approaches in the treatment of PTSD. *PTSD Res Q*. 2017;28(2):1050-1835. https://www.ptsd.va.gov/professional/newsletters/research-quarterly/V28N2.pdf.

- 19. Engel GL. The need for a new medical model: A challenge for biomedicine. *Science* (80-). 1977;196(4286):129-136.
- 20. Friedmann E, Son H, Salem M. The animal-human bond: Health and wellness. In: Fine AH, ed. *Handbook on Animal Assisted Therapy, Theoretical Foundations and Guidelines for Practice*. 4th ed. Burlington, MA: Academic Press; 2015:73-90.
- 21. Yehuda R. Post-traumatic stress disorder. *N Engl J Med*. 2002;356(2):108-114. doi:10.1056/NEJMra012941.
- 22. Yount R, Ritchie E, Laurent MS, Chumley P, Olmert M. The role of service dog training in the treatment of combat-related PTSD. *Psychiatr Ann.* 2013;43:292-295. doi:10.3928/00485713-20130605-11.
- 23. Fine AH. *Handbook on Animal-Assisted Therapy: Foundations and Guidelines for Animal-Assisted Interventions*. 4th ed. Academic Press; 2015.
- 24. Sherin JE, Nemeroff CB. Post-traumatic stress disorder: The neurobiological impact of psychological trauma. *Dialogues Clin Neurosci.* 2011;13(3):263-278.
- 25. Boscarino JA. Psychobiologic predictors of disease mortality after psychological trauma: implications for research and clinical surveillance. *J Nerv Ment Dis.* 2008;196(2):100-107. doi:10.1097/NMD.obo13e318162a9f5.
- 26. Elzinga BM, Schmahl CG, Vermetten E, van Dyck R, Bremner JD. Higher cortisol levels following exposure to traumatic reminders in abuse-related PTSD. *Neuropsychopharmacology*. 2003;28(9):1656-1665. doi:10.1038/sj.npp.1300226.
- 27. Thoma MV, Joksimovic L, Kirschbaum C, Wolf JM, Rohleder N. Altered salivary alpha-amylase awakening response in Bosnian War refugees with posttraumatic stress disorder. *Psychoneuroendocrinology*. 2012;37(6):810-817. doi:10.1016/j.psyneuen.2011.09.013.
- 28. Fink G. Stress of War, Conflict and Disaster. Oxford, UK: Academic Press; 2010.
- 29. Rohleder N, Nater UM, Wolf JM, Ehlert U, Kirschbaum C. Psychosocial stress-induced activation of salivary alpha-amylase: An indicator of sympathetic activity? *Ann N Y Acad Sci.* 2004;1032(1):258-263. doi:10.1196/annals.1314.033.
- 30. Kang Y. Psychological stress-induced changes in salivary alpha-amylase and adrenergic activity. *Nurs Heal Sci.* 2010;12(4):477-484. doi:10.1111/j.1442-2018.2010.00562.x.
- 31. Tan G, Dao TK, Farmer L, Sutherland RJ, Gevirtz R. Heart rate variability (HRV) and posttraumatic stress disorder (PTSD): A pilot study. *Appl Psychophysiol Biofeedback*. 2011;36(1):27-35. doi:10.1007/s10484-010-9141-y.
- 32. Friedmann E, Thomas SA, Stein PK, Kleiger RE. Relation between pet ownership and heart rate variability in patients with healed myocardial infarcts. *Am J Cardiol*. 2003;91(6):718-721.
- 33. Friedmann E, Son H. The human-companion animal bond: How humans benefit. *Vet Clin North Am Small Anim Pract*. 2009;39(2):293-326. doi:10.1016/j.cvsm.2008.10.015.
- 34. Barker SB, Knisely JS, McCain NL, Schubert CM, Pandurangi AK. Exploratory study of stress-buffering response patterns from interaction with a therapy dog. *Anthrozoos*. 2010;23(1):79-91. doi:10.2752/175303710X12627079939341.
- 35. Duncan S. PAWS Program Effectiveness Analysis- Q20. Lubbock, TX: Quan-Qual Outcomes; 2011.
- 36. Furst G. Animal Programs in Prison: A Comprehensive Assessment. Lynee Rienner Publishers; 2011.
- 37. Mulcahy C. Companions on the inside: Pet ownership and the introduction of a prison dog program at Darling Downs Correctional Centre (unpublished master's thesis). 2011.
- 38. Richardson-Taylor K, Blanchette K. *Results of an Evaluation of the Pawsitive Directions Canine Program at Nova Institution for Women*. Ottawa, Ontario; 2001. http://www.csc-scc.gc.ca/research/092/r108\_e.pdf.

- 39. Pedersen I, Nordaunet T, Martinsen EW, Berget B, Braastad BO. Farm animal-assisted intervention: relationship between work and contact with farm animals and change in depression, anxiety, and self-efficacy among persons with clinical depression. *Issues Ment Heal Nurs*. 2011;32(8):493-500. doi:10.3109/01612840.2011.566982.
- 40. Souter MA, Miller MD. Do animal-assisted activities effectively treat depression? A meta-analysis. *Anthrozoos*. 2007;23(1):7-19. doi:10.2752/175303707X207954.
- 41. Barker SB, Dawson KS. The effects of animal-assisted therapy on anxiety ratings of hospitalized psychiatric patients. *Psychiatr Serv.* 1998;49(6):797-801. doi:10.1176/ps.49.6.797.
- 42. Nordgren L, Engstrom G. Animal-assisted intervention in dementia: Effects on quality of life. *Clin Nurs Res.* 2014;23(1):7-19. doi:10.1177/1054773813492546.
- 43. Bernstein PL, Friedmann E, Malaspina A. Animal-assisted therapy enhances resident social interaction and initiation in long-term care facilities. *Anthrozoos*. 2000;13(4):213-224. doi:10.2752/089279300786999743.
- 44. Krause-Parello CA, Morales KA. Military veterans and service dogs: A qualitative inquiry using interpretive phenomenological analysis. *Anthrozoos*. 2018;31(1):61-75. doi:10.1080/08927936.2018.1406201.
- 45. Laffaye C, Cavella S, Drescher K, Rosen C. Relationships among PTSD symptoms, social support, and support source in veterans with chronic PTSD. *J Trauma Stress*. 2008;21(4):394-401. doi:10.1002/jts.20348.
- 46. Meadows LA, Kaslow NJ, Thompson MP, Jurkovic GJ. Protective factors against suicide attempt risk among African American women experiencing intimate partner violence. *Am J Community Psychol* . 2005;36(1-2):109-121. doi:10.1007/s10464-005-6236-3.
- 47. Compton MT, Thompson NJ, Kaslow NJ. Social environment factors associated with suicide attempt among low- income African Americans: The protective role of family relationships and social support. *Soc Psychiatry Psychiatr Epidemiol.* 2005;40(3):175-185. doi:10.1007/s00127-005-0865-6.
- 48. Post SG. It's good to be good: 2011 fifth annual scientific report on health, happiness and helping others. *Int J Pers Cent Med.* 2011;1(4):814-829. doi:10.5750/IJPCM.V1I4.154.
- 49. Schwartz C, Meisenhelder JB, Ma Y, Reed G. Altruistic social interest behaviors are associated with better mental health. *Psychosom Med.* 2003;65(5):778-785.
- 50. Montpetit AJ, Alhareeri AA, Montpetit M, et al. Telomere length: A review of methods for measurement. *Nurs Res.* 2014;63(4):289-299. doi:10.1097/NNR.00000000000037.
- 51. Axelrad MD, Budagov T, Atzmon G. Telomere length and telomerase activity; A yin and yang of cell senescence. *J Vis Exp.* 2013;75:e50246. doi:10.3791/50246.
- 52. Darrow SM, Verhoeven JE, Revesz D, et al. The association between psychiatric disorders and telomere length: A meta-analysis involving 14,827 persons. *Psychosom Med* . 2016;78(7):776-787. doi:10.1097/PSY.00000000000356.
- 53. Zhang L, Hu XZ, Benedek DM, et al. The interaction between stressful life events and leukocyte telomere length is associated with PTSD. *Mol Psychiatry*. 2014;19(8):855-856. doi:10.1038/mp.2013.141.
- 54. Ladwig KH, Brockhaus AC, Baumert J, et al. Posttraumatic stress disorder and not depression is associated with shorter leukocyte telomere length: findings from 3,000 participants in the population-based KORA F4 study. *PLoS One*. 2013;8(7):e64762. doi:10.1371/journal.pone.0064762.
- 55. Epel E. How "reversible" is telomeric aging? *Cancer Prev Res.* 2012;5(10):1163-1168. doi:10.1158/1940-6207.CAPR-12-0370.
- 56. Ornish D, Lin J, Daubenmier J, et al. Increased telomerase activity and comprehensive lifestyle changes: A pilot study. *Lancet Oncol.* 2008;9(11):1048-1057. doi:10.1016/S1470-2045(08)70234-1.
- 57. Boks MP, van Mierlo HC, Rutten BP, et al. Longitudinal changes of telomere length and epigenetic age

- related to traumatic stress and post-traumatic stress disorder. *Psychoneuroendocrinology*. 2015;51:506-512. doi:10.1016/j.psyneuen.2014.07.011.
- 58. Zenithson N, Albright J, Fine A, Peralta J. Our ethical and moral responsibility: Ensuring the welfare of therapy animals. In: Fine AH, ed. ). *Handbook on Animal-Assisted Therapy: Foundations and Guidelines for Animal-Assisted Interventions*. 4th ed. California: Elsevier; 2015.
- 59. Bergamasco L, Osella MC, Savarion P, et al. Heart rate variability and saliva cortisol assessment in shelter dog: Human-animal interaction effects. *Appl Anim Behav Sci.* 2010;125(1-2):56-68. doi:10.1016/j.applanim.2010.03.002.
- 60. Glenk LM. Current perspectives on therapy dog welfare in animal-assisted interventions. *Animals*. 2017;7(2):7. doi:10.3390/ani7020007.
- 61. Bowen DJ, Kreuter M, Spring B, et al. How we design feasibility studies. *Am J Prev Med.* 2009;36(5):452-457. doi:10.1016/j.amepre.2009.02.002.
- 62. Krause-Parello CA, Levy C, Holman E, Kolassa JE. Effects of VA facility dog on hospitalized veterans seen by a palliative care psychologist: An innovative approach to impacting stress indicators. *Am J Hosp Palliat Med.* 2018;35(1):5-14. doi:10.1177/1049909116675571.
- 63. Krause-Parello, C A, Tychowski J, Gonzalez A, Boyd Z. Human-canine interaction: Exploring stress indicator response patterns of salivary cortisol and immunoglobulin A. *Res Theory Nurs Pr*. 2012;26(1):25-40.
- 64. Gee NR, Friedmann E. Heart rate variability during a working memory task: Does touching a dog or person affect the response? *Anthrozoos*. 2014;27(4):513-526. doi:10.2752/089279314X14072268687763.
- 65. Krause-Parello C, Friedmann E. The use of animal-assisted intervention to examine the effects of salivary alpha-amylase, immunoglobulin A, and heart rate during forensic interviews in child sexual abuse cases. *Anthrozoos*. 2014;27(4):582-590. doi:10.2752/089279314X14072268688005.
- 66. Alvarez JR, Yount RA, Puckett M, Wyman C, McLean C MS. Implementation and effectiveness of an assistance dog training intervention for PTSD. In: Baltimore, MD: The Veterans Administration Mental Health Conference; 2009.
- 67. United States Census Bureau. QuickFacts: Montgomery County, Maryland. https://www.census.gov/quickfacts/fact/table/montgomerycountymaryland/VET605216#viewtop.
- 68. Yount RA, Olmert MD, Lee MR. Service dog training program for treatment of posttraumatic stress in service members. *US Army Med Dep J.* 2012:63-69.
- 69. Furukawa TA, Noma H, Caldwell DM, et al. Waiting list may be a nocebo condition in psychotherapy trials: A contribution from network meta-analysis. *Acta Psychiatr Scand*. 2014;130(3):181-192. doi:10.1111/acps.12275.
- 70. Weathers FW, Litz BT, Keane TM, Palmieri PA, Marx BP, Schnurr PP. The PTSD Checklist for DSM-5 (PCL-5). 2013. http://www.ptsd.va.gov/professional/assessment/adult-sr/ptsd-checklist.asp.
- 71. Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The posttraumatic stress disorder checklist for DSM-5 (PCL-5): Development and Initial psychometric evaluation. *J Trauma Stress*. 2015;28(6):489-498. doi:10.1002/jts.22059.
- 72. PROMIS. NIH Toolbox Perceived Stress Fixed Form Age 18+ v2.0. 2018. http://www.healthmeasures.net/index.php?option=com\_instruments&view=measure&id=683&Itemid=992.
- 73. Salsman JM, Butt Z, Pilkonis PA, et al. Emotion assessment using the NIH Toolbox. *Neurology*. 2013;80(11 Suppl 3):S76-86. doi:10.1212/WNL.obo13e3182872e11.
- 74. PROMIS. Validation. 2018. http://www.healthmeasures.net/explore-measurement-systems/promis/measure-development-research/validation.

- 75. PROMIS. PROMIS Short Form v1.0 Positive Affect 15a. 2017. http://www.healthmeasures.net/index.php?option=com\_instruments&view=measure&id=835&Itemid=992.
- 76. Iqbal SU, Rogers W, Selim A, et al. The Veterans RAND 12 item health survey (VR-12): What it is and how it is used. 2007. http://www.hosonline.org/globalassets/hosonline/publications/veterans\_rand\_12\_item\_health\_survey\_vr-12\_2007.pdf.
- 77. Chum A, Skosireva A, Tobon J, Hwang S. Construct validity of the SF-12v2 for the homeless population with mental illness: An Instrument to measure self-reported Mental and physical health. *PLoS One*. 2016;11(3):e0148856. doi:10.1371/journal.pone.0148856.
- 78. Campbell-Sills L, Stein MB. Psychometric analysis and refinement of the Connor-davidson Resilience Scale (CD-RISC): Validation of a 10-item measure of resilience. *J Trauma Stress*. 2007;20(6):1019-1028. doi:10.1002/jts.20271.
- 79. Griffin DW, Bartholomew K. The metaphysics of measurement: The case of adult attachment. In: *Advances in Personal Relationships, Vol 5. Attachment Processes in Adulthood.* London, England: Jessica Kingsley Publishers; 1994:17-52.
- 80. PROMIS PROMIS Short Form v2.0 Satisfaction with Social Roles and Activities 4a. 2018. http://www.healthmeasures.net/index.php?option=com\_instruments&view=measure&id=206&Itemid=992.
- 81. Bartlett SJ, Orbai AM, Duncan T, et al. Reliability and validity of selected PROMIS measures in people with Rheumatoid Arthritis. *PLoS One*. 2015;10(9):e0138543. doi:10.1371/journal.pone.0138543.
- 82. Nagl M, Gramm L, Heyduck K, Glattacker M, Farin E. Development and psychometric evaluation of a German version of the PROMIS® item banks for satisfaction with participation. *Eval Health Prof.* 2015;38(2):160-180. doi:10.1177/0163278713503468.
- 83. PROMIS. PROMIS Short Form v1.0 Satisfaction with Participation in Discretionary Social Activities 7a. 2018. http://www.healthmeasures.net/index.php?option=com\_instruments&view=measure&id=176&Itemid=992.
- 84. PROMIS PROMIS Short Form v2.0 Companionship 4a. 2018. doi:http://www.healthmeasures.net/index.php?option=com\_instruments&view=measure&id=195&Ite mid=992.
- 85. Hahn EA, DeWalt DA, Bode RK, et al. New English and Spanish social health measures will facilitate evaluating health determinants. *Heal Psychol.* 2014;33(5):490-499. doi:10.1037/hea0000055.
- 86. PROMIS. PROMIS Short Form v1.0 Depression 8a (PROMIS-D). 2017. http://www.healthmeasures.net/index.php?option=com\_instruments&view=measure&id=156&Itemid=992.
- 87. Pilkonis P.A., Yu L, Dodds NE, Johnston KL, Maihoefer CC, Lawrence SM. Validation of the depression item bank from the Patient-Reported Outcomes Measurement Information System (PROMIS®) in a three-month observational study. *J Psychiatr Res.* 2014;56:112-119. doi:10.1016/j.jpsychires.2014.05.010.
- 88. Schalet BD, Cook K.F., Choi SW, Cella D. Establishing a common metric for self-reported anxiety: Linking the MASQ, PANAS, and GAD-7 to PROMIS anxiety. *J Anxiety Disord*. 2014;28(1):88-96. doi:10.1016/j.janxdis.2013.11.006.
- 89. Beck AT, Kovacs M, Weissman A. Assessment of suicidal intention: the Scale for Suicide Ideation. *J Consult Clin Psychol.* 1979;47(2):343-352.
- 90. O'Callaghan NJ, Varinderpal DS, Thomas P, Fenech M. A quantitative real-time PCR method for absolute telomere length. *Biotechniques*. 2008;44(6):807-809. doi:10.2144/000112761.
- 91. Gácsi M, Maros K, Sernkvist S, Faragó T, Miklósi Á. Human analogue safe haven effect of the owner:

- Behavioural and heart rate response to stressful social stimuli in dogs. *PLoS One*. 2013;8(3):e58475. doi:10.1371/journal.pone.0058475.
- 92. Son H, Friedmann E, Thomas SA. Application of pattern mixture models to address missing data in longitudinal data analysis using SPSS. *Nurs Res.* 2012;61:195-203. doi:10.1097/NNR.ob013e3182541d8c.
- 93. Hanisch SE, Twomey CD, Szeto ACH, Birner UW, Nowak D, Sabariego C. The effectiveness of interventions targeting the stigma of mental illness at the workplace: A systematic review. *BMC Psychiatry*. 2016;16(1). doi:10.1186/s12888-015-0706-4.
- 94. Sin NL, Lyubomirsky S. Enhancing well-being and alleviating depressive symptoms with positive psychology interventions: A practice-friendly meta-analysis. *J Clin Psychiatry*. 2009;65(5):467-487. doi:10.1002/jclp.20593.